CLINICAL TRIAL: NCT04946890
Title: Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Effectiveness of MRX2843 Tablets in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Study of MRX2843 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-66M12
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Acute Myeloid Leukemia Leukemia
Keywords: MRX2843
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — MRX-2843

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MRX2843 orally 80 mg/d (Experimental): Participants received 80 mg MRX2843 administered orally (PO), once daily (QD), in a fasted state on Days
  1 to 21 of a 21-day cycle.
  Interventions: Drug: MRX2843
- MRX2843 orally 120 mg/d (Experimental): Participants received 120 mg MRX2843 administered orally (PO), once daily (QD), in a fasted state on Days
  1 to 21 of a 21-day cycle.
  Interventions: Drug: MRX2843
- MRX2843 orally 180 mg/d (Experimental): Participants received 180 mg MRX2843 administered orally (PO), once daily (QD), in a fasted state on Days
  1 to 21 of a 21-day cycle.
  Interventions: Drug: MRX2843

INTERVENTIONS:
Drug: MRX2843 — MRX2843 is treated at 80mg/d, 120mg/d and 180mg/d respectively

SUMMARY:
Patients will receive oral MRX2843 for 28 days to study the side effects, tolerability and best dose for treating relapsed or refractory acute myeloid leukemia With FLT3 Mutations.

DETAILED DESCRIPTION:
It is open-label, dose escalation study designed to characterize the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of orally administered MRX2843 as a single agent given daily for 28 days.

The study includes two parts, Phase I and Phase II, and is carried out in three phases. The Phase I clinical study is divided into two phases: the dose escalation study (Ia) and the expanded enrollment study (Ib). The third phase is the phase II research phase, which is designed based on phase I clinical results.

Phase Ia：Cohorts of 3 patients receive MRX2843 until dose limiting toxicity is noted (DLT). At that point cohorts will expand to 6 patients until MTD is determined.

Phase Ib/ II：According to the relevant data on safety and effectiveness, expand the enrollment of FLT3 mutation relapsed/refractory AML patients at the appropriate dose

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥ 18 years;
2. Expected survival period ≥ 12 weeks;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. Histopathologically documented primary or secondary AML, as defined by WHO criteria, confirmed by pathology review at treating institution, meeting at least one of the following: i. After complete remission, leukemia cells reappear in peripheral blood, or the ratio of bone marrow immature cells to bone marrow cells> 5%, or leukemia cell infiltration outside the bone marrow; ii. After standard protocol (including cytarabine and a kind of Anthracycline or anthraquinone drugs) for refractory AML patients who have not achieved complete remission after two courses of treatment;
5. During the dose escalation phase, there is no need to test for FLT3 mutation status; for the expansion of the enrollment and phase II study phase, the FLT3 mutation status test results within the past 6 months will be accepted; if not, the central laboratory or research center needs to test and confirm the test Patients with FLT3 mutation status in bone marrow or whole blood. The test results show that the subject has any of the following FLT3 mutation types, and can be included in the group: FLT3 internal tandem repeat (ITD), FLT3 tyrosine kinase domain (TKD);
6. Laboratory inspection must meet the following standards:

   1. Blood routine: Under normal circumstances, the white blood cell count (WBC) ≤20×109/L; or the patient's white blood cell count (WBC)>20×109/L before using hydroxyurea or cytarabine, use for a period of time and stop the drug After 3 days, check the white blood cell count (WBC) ≤20×109/L;
   2. Blood coagulation function: the international standardized ratio of prothrombin time and partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN);
   3. Liver: If there is no clear liver metastasis, serum total bilirubin ≤1.5 ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN; if there is clear Gilbert syndrome (Unconjugated hyperbilirubinemia), total bilirubin ≤ 3.0 ULN;
   4. Kidney: Serum creatinine (Scr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥50 mL/min (calculated according to Cockcroft-Gault formula);
7. Normal or abnormal ocular retinal examination has no clinical significance;

Exclusion Criteria:

1. Previously received medications targeting MerTK and/or FLT3
2. Histologic diagnosis of acute promyelocytic leukemia;
3. Have had other malignant tumors in the past 5 years ;
4. Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher;
5. The tumor involves the central nervous system and/or the testis;
6. Active, uncontrolled infection;
7. Radiation therapy within 4 weeks prior to study;
8. Received systemic glucocorticoids within 14 days before the first dose ；
9. Left ventricular ejection fraction ≤1 × ULN,or﹤50%. Clinically significant ECG QTc prolongation (Male: >450ms, Female: >470ms).Significant cardiac disease；
10. Human immunodeficiency virus positivity;
11. Active hepatitis B or C or other active liver disease;
12. Women who are pregnant, lactating;
13. Have a history or family history of known or suspected retinitis pigmentosa;
14. Inability to swallow drugs orally, and conditions that seriously affect the absorption or pharmacokinetic parameters of the test drug;
15. History of type 1 diabetes;
16. Any situation that is unstable or may endanger the safety of patients and their compliance with research;
17. Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize patient safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 Days
  Safety: Incidence of dose limiting toxicity (DLT)and Adverse Event (AE)
RP2D | 28 Days
  Explore the maximum tolerated dose (MTD) and phase II recommended dose (RP2D), and initially formulate a reasonable dosing plan;

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 28 Days
  Maximum serum concentration (Cmax)
Area under the plasma concentration-time curve (AUC) from time zero to the time point of t (AUC0-tn) | 28 Days
  Area under the plasma concentration-time curve (AUC) from time zero to the time point of t (AUC0-tn)
Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-inf) | 28 Days
  Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-inf)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 28 Days
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Apparent volume of distribution at equilibrium after oral administration（Vss/F） | 28 Days
  Apparent volume of distribution at equilibrium after oral administration（Vss/F）
Plasma Decay Half-Life (t1/2z) | 28 Days
  Plasma Decay Half-Life (t1/2z)
Apparent Oral Clearance (CLz/F) | 28 Days
  Apparent Oral Clearance (CLz/F)
Average plasma or serum concentration(Cav) | 28 Days
  Average plasma or serum concentration(Cav)
changes in FLT3 mutation status in plasma | 28 Days
  changes in FLT3 mutation status in plasma
Rate of Complete Remission (CR) | 28 Days
  Rate of Complete Remission (CR)
Rate of partial remission (PR) | 28 Days
  Rate of partial remission (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Junmin Li，Ph.D, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No